CLINICAL TRIAL: NCT06722040
Title: Effect and Safety of Implementing a Pediatric Triage Track in a Public Medical Helpline in Denmark
Brief Title: Effect and Safety of a Pediatric Triage Track on Hospital Visits and at the Public Medical Helpline 1813, Capital Region, Denmark
Status: Completed | Type: Observational
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Responsible Party: Sponsor
Other Study IDs: EMSCRDenmark
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Emergency Medical Services; Telemedicine; Children; Triage; Hospital Admission
Keywords: Pediatric Triage track; MH1813; Medical Helpline 1813; EMS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before pediatric triage track: The dyads of children and their caregivers calling the Medical Helpline 1813 before the implementation of the pediatric triage unit (January 1, 2022 - June 30, 2022)
- After pediatric Triage track: The dyads of children and their caregivers calling the Medical Helpline 1813 after the implementation of the pediatric triage unit (January 1, 2023-June 30, 2023)
  Interventions: Other: Implementation of a pediatric triage track

INTERVENTIONS:
Other: Implementation of a pediatric triage track — In 2023, a pediatric triage track was implemented at MH1813 to route calls concerning children to specialists in pediatrics, ensuring better expertise.
  Groups: After pediatric Triage track

SUMMARY:
Children under three years old often fall ill. While most illnesses are mild, they often lead to worry which contributes to a high number of contacts with general practitioners and acute medical services such as the Medical Helpline 1813 (MH1813). The MH1813 is a free urgent medical helpline staffed by healthcare professionals and intended for acute medical conditions that cannot wait until the general practitioner is available the following day. About 25% of the calls to MH1813 regards a child under the age of 10 years. To improve triage, MH1813 implemented video triage and educational video tutorials for parents. In July 2022, a pediatric triage track was established to route calls concerning children to specialists in pediatrics, ensuring better expertise. The hypothesis is that this new pediatric triage track have reduced hospital referrals safely, without increasing ambulance dispatches or severe incidents.

DETAILED DESCRIPTION:
Background Children below the age of three experience on average three sick days per month, leading to their absence from daycare centers.(1) Fortunately, young children most often have mild symptoms and do not require medical interventions or physical evaluation by a doctor. However, parents of sick children report significant worry,(2,3) which may explain the high number of acute contacts with general practitioners, the MH 1813 and other out-of-hours medical services, as well as hospital referrals.

The Medical Helpline 1813

The MMH1813, Copenhagen Medical Services, Capital Region, serves 1.8 million citizens, including 240,000 under 12 years. The MH1813 is staffed by nurses and physicians. The call-handler has two options at the end of the call:

1. Patient self-care at home, with the option to repeat the contact to the MH1813 or contact the general practitioner the following day, or
2. refer the patient to hospitals in the Capital Region, Denmark.

In 2021, the MH1813 received about 1 million calls, and close to 25% involved children aged 0-10 years.(4) The quality of telephone triage at the MH1813 greatly impacts affected children, parents, and the healthcare system. Similar services are used in other countries and are expected to be implemented in other regions of Denmark in the future.

Telephone triage of children Correct and optimal triage of ill children is a huge challenge across the healthcare system. The parents are typically concerned about their child, and the description of the child's symptoms, essential for correct triage, relies solely on the parent.(2) Data from the MH1813 revealed that 16% of the parents repeated the call to the MH1813 within 72 hours, with some seeking telephone triage up to 5 times.5 Additionally, about 40% of the children were referred to a hospital, but around 40% of these children did not receive paraclinical tests or treatment besides paracetamol.(5)

The MH1813 has implemented different ways to improve telephone triage of children:

* "Video triage of children", enabling the nurse or physician to perform a triage with video of the child, complementing the information provided by the parents.(2,6,7)
* "Tips from Pediatricians". Short informative videos on the most common symptoms in ill children, guiding parents on what can be done at home and when to seek medical help.(5,8) (https://www.regionh.dk/boernelaegernesboernetips/english/Sider/default.aspx)

Implementation of a pediatric triage track Before July 2022, calls regarding children to MH1813 received triage by the first available nurse or physician regardless of their level of expertise in pediatric triage. In July 2022 a pediatric triage track was implemented, directing calls regarding children less than 12 years old to a team of healthcare professionals with specialized clinical experience in pediatrics. This team consists of nurses, general practitioners, pediatricians, or doctors in training to be pediatricians. By the 1st of November 2022, all members of the pediatric triage track had received training in telephone triage for children and spent a day assisting in triaging children at a pediatric department at a hospital. Furthermore, by April 11, 2023, the MH1813 established a pediatric consultant during the peak hours on weekdays (5 pm - 10 pm). The pediatric consultant was either a pediatrician or a doctor in training to be a pediatrician with a current affiliation with a pediatric department at a hospital. As a part of the triage process of children at the MH1813, all referrals of to the hospital should be discussed with the pediatric consultant by the call-handlers.

Hypothesis We hypothesize that the introduction of a pediatric triage track results in a reduced proportion of children referred to hospitals during the primary call and that it is safe. Safety will be defined by no increase in the proportion of dispatched ambulances within 72 hours from the primary call, or in the proportion of children admitted to the Intensive Care Unit, or in the proportion of reports from the hospitals regarding children with serious accidental incidents after telephone triage at the MH1813.

Aim To analyze whether the implemented pediatric triage track contributes to decreasing the proportion of children examined at hospitals and, secondary, a decrease in the proportion of parents who repeat the call to MH1813 for telephone triage, and that it is safe.

Method Design: A register-based cohort study. Before telephone triage, callers are asked to enter the Civil Registration Number for the individual the call refers to, from which the age is electronically calculated.

The two exposure groups are:

* The dyads of children and their caregivers calling the Medical Helpline 1813 before the introduction of the pediatric triage unit (January 1, 2022 - June 30, 2022)
* The dyads of children and their caregivers calling the Medical Helpline 1813 after the introduction of the pediatric triage unit (January 1, 2023-June 30, 2023)

Setting: The MH1813, Copenhagen Medical Services, Capital Region, Denmark, the Departments of Paediatrics and Adolescent Medicine in the Capital Region, and the general practitioners in the Capital Region.

Participants: Children in the Capital Region younger than 12 years (about 244,000), and their parents (approximately 488,000).

Statistical analysis and data management The MH1813 receives about 250,000 calls annually regarding children under 12 years. We will compare all calls regarding children under 12 years for the two periods with around 125,000 children in each group.

We will collect the following information from administrative data at the MH1813, Copenhagen Emergency Services: Civil Registration Number, sex, age of the child, date of call, call duration, the profession of the call handler (nurse/physician) during the primary call, actions during the telephone triage (use of video triage, use of Tips from pediatricians, referral to self-care or hospital).

We will also collect information on of repeated calls for telephone triage within 72 hours from the primary call, and dispatch of ambulances from the Copenhagen Emergency Services within 72 hours from the primary call.

We will use the civil registration number to collect further information from national health registers: The Danish National Patient Register: Registered date, time, and diagnoses for (admission and) discharge from the hospitals 12 hours prior to 72 hours after the primary call to MH1813. Similarly, we will collect information on all admissions to an intensive care unit 12 hours prior to 72 hours after the primary call to MH1813.

The Danish National Health Services Register: Number and types (e-mail, telephone, physical examination) of contacts to the general practitioner within 72 hours after the primary call.

All analyses will be done in R version 3.6.0.

Power analysis The primary outcome of our study is the change in the proportion of children referred to hospitals from MH1813 after the primary call. To detect a 1%-point decrease from the current 40% to 39%, we need to include 105,536 dyads of children and caregivers calling the MH 1813, to achieve a power of 90%, with a two-sided test, and a 95% confidence level. To detect a 5%-point decrease, from 40% to 35%, we need to include 4,048 dyads.

Ethical considerations and approvals This is a prospective register-based study and ethical approval is not required for these studies in Denmark. The project will be registered at the Capital Region at Knowledge Center for Data reviews, Privacy. All personal data will be stored according to the Danish GPDR rules in a secured encrypted server with limited logged access. Data will be stored for 10 years.

Perspectives Investigating strategies to improve telephone triage of children holds significant relevance to the primary, hospital, and prehospital sectors in Denmark. It has a great impact on a substantial population - children and their parents. The MH1813 handles 250,000 contacts each year regarding children, and similar out-of-hours solutions are poised for implementation in other regions of the country.

In the Capital Region, 40% of sick children referred to hospitals did not need treatment or paraclinical examinations.(5) Many of these cases could have been effectively managed at home by their parents, eliminating the need for hospital visits and associated waiting times. Actions to ensure better telephone triage will result in fewer children with mild symptoms at the hospitals and enable a more strategic use of resources in the health system. We expect our findings, to be useful across the health sectors in Denmark to all regions of Denmark, and other countries, and inspire solutions for other patient groups.

Behind the project The project will originate from a collaboration between the Emergency Medical Services, Capital Region, Denmark, a part of the prehospital sector, the Departments of Pediatrics and Adolescent Medicine, both at the Copenhagen University Hospital Hvidovre, Denmark, and the Copenhagen University Hospital Herlev, Denmark.

References

1. Pönkä, A., Nurmi, T., Salminen, E. & Nykyri, E. Infections and other illnesses of children in day-care centers in Helsinki I: Incidences and effects of home and day-care center variables. Infection 19, 230-236 (1991).
2. Gren, C. et al. How parents express their worry in calls to a medical helpline: a mixed methods study. BMC primary care 23, 80 (2022).
3. Uldall, P. Spæd- Og Småbørns Almindelige Sygelighed - Forekomst Og Sociale Konsekvenser. (Fadl's Forlag, København, 1987).
4. Rasmussen, M. Section for data, controlling and IT, Copenhagen Emergency Centre. (2019).
5. Borch-Johnsen, L. et al. Video Tutorials to Empower Caregivers of Ill Children and Reduce Health Care Utilization: A Randomized Clinical Trial. JAMA Netw Open 6, e2336836-e2336836 (2023).
6. Gren, C. et al. 'We can't do without it': Parent and call-handler experiences of video triage of children at a medical helpline. PLoS One 17, e0266007 (2022).
7. Gren, C. et al. Video triage of children with respiratory symptoms at a medical helpline is safe and feasible-a prospective quality improvement study. PLoS One 18, e0284557 (2023).
8. Borch-Johnsen, L. et al. Development of video tutorials to help parents manage children with acute illnesses using a modified Delphi method. Acta Paediatr 112, 1574-1585 (2023).

ELIGIBILITY:
Inclusion Criteria:

Calls regarding children aged up to 11.9 years

Exclusion Criteria:

Calls regarding children or adults older than 12 years

Ages: 0 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children in the Capital Region younger than 12 years
Sampling Method: Probability Sample
Enrollment: 244000 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Referral to hospital after the primary call to Medical Helpline 1813 (MH1813) | 72 hours from the primary call to MH1813

SECONDARY OUTCOMES:
Duration of the primary call | During the primary call to MH1813
Children referred to hospitals within 72 hours after the primary call | 72 hours from the primary call to MH1813
Children who received video triage during the primary call | During the primary call to MH1813
"Tips from Pediatricians" sent to parents during the primary call | During the primary call to MH1813
Repeated calls for telephone triage within 72 hours from the primary call | 72 hours from the primary call to MH1813
Children examined at hospitals within 72 hours after the primary call | 72 hours from the primary call to MH1813
Duration of hospital admission and admission lengths: 0-11.9 hours, 12-23.9 hours, 24-72 hours, more than 72 hours | 72 hours from the primary call to MH1813
Hospital discharge diagnoses within 72 hours after the primary call | 72 hours from the primary call to MH1813
Children examined at hospital with diagnoses related to mild diseases | 72 hours from the primary call to MH1813

OTHER OUTCOMES:
Severe adverse outcomes: | 72 hours from the primary call to MH1813
  Dispatched ambulances from the MH1813 within 72 hours from the primary call. Children admitted to the intensive care unit within 72 hours after the primary call.
  Reports from the hospitals to the MH1813 regarding children with serious adverse event within 72 hours after primary telephone triage at the MH1813.
  Children admitted to hospitals with diagnoses related to severe diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Medical Services Capital Region, Denmark, Ballerup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided